CLINICAL TRIAL: NCT03300726
Title: Cerebrospinal Fluid Markers of Synaptic Injury and Functional Connectivity in Alzheimer's Disease
Brief Title: Synaptic Injury and Functional Connectivity in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Rawan Tarawneh, Assistant Professor of Neurology, Ohio State University
Other Study IDs: 2017H0255
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease, Late Onset
Keywords: Synaptic injury
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Cerebrospinal fluid (CSF) and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCI due to AD or mild AD dementia: The clinical diagnoses of amnestic MCI due to AD or mild AD dementia will be made according to standard clinical criteria as described by the National Institute of Aging -Alzheimer's Association Working Group and supported by CSF biomarker data for tau, p-tau181, and Aβ42. This includes evaluation for other systemic or neurological disorders which could account for the cognitive impairment, and inclusion of results from ancillary structural imaging (CT or structural MRI), neuro-psychometric testing, and FDG-PET imaging (when available) into the diagnostic scheme. All participants in this group will undergo clinical and cognitive evaluations, CSF analysis, and functional MRI during resting state and semantic memory tasks.
  Interventions: Diagnostic Test: CSF analysis; Radiation: Functional MRI
- Normal controls: Normal cognition will be defined as cognitive performance on detailed neuropsychometric testing that falls within 1 SD of age-, gender-, and education-matched norms in all cognitive domains, and no subjective report of cognitive decline from an individual's baseline (i.e. CDR 0). All participants in this group will undergo clinical and cognitive evaluations, CSF analysis, and functional MRI during resting state and semantic memory tasks.
  Interventions: Diagnostic Test: CSF analysis; Radiation: Functional MRI

INTERVENTIONS:
Diagnostic Test: CSF analysis — CSF analysis for tau, p-tau181, Abeta42, and CSF levels of markers of synaptic injury
Radiation: Functional MRI — Functional MRI during resting state and semantic memory task activation

SUMMARY:
The purpose of this study is to examine cross-sectional associations between CSF markers of synaptic injury (Ng and SNAP-25) and functional connectivity in default and semantic memory networks using 3T- fMRI in individuals with MCI (i.e. the earliest clinically detectable stage of cognitive impairment) due to AD or mild AD dementia (CDR 0.5-1; n=20) and cognitively normal controls (CDR 0; n=20).

DETAILED DESCRIPTION:
SPECIFIC AIMS:

Aim 1: Investigate correlations between CSF biomarkers of synaptic injury (Ng and SNAP-25) and functional connectivity (FC) within the default mode network (DMN) using resting-state fMRI (adjusting for age, gender, apolipoprotein-E4 [APOE4] genotype, task performance, and regional brain atrophy) in MCI/AD and controls.

Aim 2: Examine correlations between CSF biomarkers of synaptic injury and functional connectivity (FC) within the semantic memory network on task-activated fMRI using the Famous Name Discrimination Task (FNDT) (adjusting for age, gender, APOE4 genotype, task performance, and regional brain atrophy) in MCI/AD and controls.

ELIGIBILITY:
Inclusion Criteria: Participants included in the study should meet all 4 inclusion criteria:

1. 60 years of age or older
2. A clinical diagnosis of MCI, mild AD dementia, or normal cognition
3. No significant medical or surgical co-morbidities
4. No contraindications to LP or MRI.

Exclusion criteria: Participants with any of the following criteria will be excluded from the study:

1. Participants with MCI due to AD or mild AD dementia who have been treated with cholinesterase inhibitors or glutamate antagonists in the 3 months prior to study enrollment
2. Individuals with any past history of ischemic or traumatic brain injury
3. Individuals with imaging evidence of significant cerebrovascular disease or structural brain lesions (e.g. tumor, demyelinating disorders, infection, or congenital anomalies)
4. Active mood disorder
5. Active alcohol use
6. Active use of benzodiazepines, barbiturates, anticholinergic, or anti-epileptic medications

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the community and the Memory Disorders Clinic of The OSU Wexner Medical Center Department of Neurology. This study will include cognitively normal individuals (CDR 0; n=20), individuals with a clinical diagnosis of single-domain or multi-domain amnestic MCI due to AD or mild AD dementia (CDR 0.5 or 1; n=20).
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Correlations between CSF biomarker measurements and fMRI measures of functional connectivity at baseline | Study duration is 3 years (36 months) for each participant, including 3 visits: one for cognitive evaluations, one for fMRI, and one for CSF collection.
  Cross-sectional associations between CSF biomarker measurements and fMRI measures at baseline

SECONDARY OUTCOMES:
CSF levels of tau, p-tau181, Abeta42, Ng, and SNAP-25 (pg/ml) | CSF collection will be performed for each participant once during the study (within 3 years of study enrollment).
  Quantification of biomarker levels in CSF
Functional Connectivity measures on functional MRI (r) | fMRI will be performed for each participant once during the study (within 3 years of study enrollment).
  Functional Connectivity Measures on fMRI during resting state and task activation

CONTACTS AND LOCATIONS:
Overall Officials: Rawan Tarawneh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No